CLINICAL TRIAL: NCT00184548
Title: A Multi-centre, Randomised, Double-blind, Parallel Group, Placebo Controlled Trial to Evaluate the Efficacy and Safety of Activated Recombinant Factor VII (rFVIIa/NovoSeven®/NiaStase®) in Severely Injured Trauma Patients With Bleeding Refractory to Standard Treatment
Brief Title: Evaluation of Recombinant Factor VIIa in Patients With Severe Bleeding
Acronym: CONTROL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F7TRAUMA-1711; 2005-002059-41 (EudraCT Number)
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Results first posted 2009-11-26 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Acquired Bleeding Disorder; Trauma
MeSH Terms: conditions — Wounds and Injuries | interventions — Factor VII

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- rFVIIa, Blunt Trauma (Experimental)
  Interventions: Drug: eptacog alfa (activated)
- Placebo, Blunt Trauma (Placebo Comparator)
  Interventions: Drug: placebo
- rVIIa, Penetrating Trauma (Experimental)
  Interventions: Drug: eptacog alfa (activated)
- Placebo, Penetrating Trauma (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: eptacog alfa (activated) — Sterile, freeze-dried powder in single-use vials to be reconstituted with sterile water for injection.
  Three doses of 200, 100 and 100 mcg/kg to be administered bolus i.v. (intravenous) over approx. three hours.
  Arms: rFVIIa, Blunt Trauma; rVIIa, Penetrating Trauma
Drug: placebo — placebo
  Arms: Placebo, Blunt Trauma; Placebo, Penetrating Trauma

SUMMARY:
This trial is conducted globally. The purpose of the trial is to evaluate that activated recombinant human factor VII (eptacog alfa (activated)) is safe and effective in severely injured trauma patients by assessing mortality and morbidity.

Please note that this trial and trial F7TRAUMA-1648 (NCT00323570) have been merged.

DETAILED DESCRIPTION:
The decision to discontinue the F7TRAUMA-1711 trial is not due to any safety concerns. The result of the pre-planned futility analysis performed in June 2008 predicted a very low likelihood of reaching a successful outcome on the primary efficacy endpoint at the end of the trial and as a consequence, the company has decided to close the trial as this juncture.

ELIGIBILITY:
Inclusion Criteria:

* Trauma injury (blunt and/or penetrating) with evidence of active hemorrhage (torso and/or proximal lower extremity) refractory to blood component therapy and surgical haemostatic procedures at the time of randomisation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 554 (Actual)
Dates: Start 2005-10; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (14):
- Novo Nordisk Clinical Trial Call Center, Princeton, New Jersey, United States
- Säo Paulo, Brazil
- Prague, Czechia
- Paris La Défense Cedex, France
- Mainz, Germany
- Vouliagment, Greece
- Kowloon, Hong Kong
- Budapest, Hungary
- Rome, Italy
- Alphen aan den Rijn, Netherlands
- Sandton, South Africa
- Madrid, Spain
- Zurich, Switzerland
- Crawley, United Kingdom

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 150 trial sites globally.
Pre-assignment Details: Eligible subjects were those with either blunt and/or penetrating trauma injuries and confirmed clinical indicators for active haemorrhage refractory to standard treatment (including blood component therapy and surgical haemostatic procedures).
Groups:
- rFVIIa, Blunt Trauma; rVIIa, Penetrating Trauma: Three single doses of activated recombinant human factor VII (rFVIIa) (200 mcg/kg, 100 mcg/kg, and 100 mcg/kg) administered over approximately three hours. First dose was administered within a maximum of 12 hours from injury. A second dose was to be administered one hour after the initial dose, and a third dose was to be administered three hours after the initial dose.
- Placebo, Blunt Trauma; Placebo, Penetrating Trauma: Three single doses of placebo (200 mcg/kg, 100 mcg/kg, and 100 mcg/kg) administered over approximately three hours. First dose was administered within a maximum of 12 hours from injury. A second dose was to be administered one hour after the initial dose, and a third dose was to be administered three hours after the initial dose.
Period: Overall Study
Arm/Group | rFVIIa, Blunt Trauma | Placebo, Blunt Trauma | rVIIa, Penetrating Trauma | Placebo, Penetrating Trauma
Started | 226 | 255 | 47 | 45
Exposed | 224 (Two subjects withdrew due to ineligibility. Excluded from safety analysis set) | 250 (Three subjects withdrew due to ineligibility, two subjects died. Excluded from safety analysis set) | 46 (One subject withdrew due to ineligibility. Excluded from safety analysis set) | 40 (Four subjects withdrew due to ineligibility, one subject died. Excluded from safety analysis set)
Completed | 218 | 242 | 44 | 38
Not Completed | 8 | 13 | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rFVIIa, Blunt Trauma | Placebo, Blunt Trauma | rFVIIa, Penetrating Trauma | Placebo, Penetrating Trauma | Total
Number analyzed (Participants) | 221 | 247 | 46 | 40 | 554
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (14.4) | 39.9 (14.2) | 33.8 (11.9) | 29.4 (10.3) | 38.4 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 65 | 3 | 3 | 130
  Male | 162 | 182 | 43 | 37 | 424

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Description: Number of participants to die from day 0 to day 30 from all causes.
Time Frame: from day 0 to 30
Population: Blunt trauma patient population: Intention-to-treat (ITT) analysis set. Patients who discontinued (withdrawn or lost to follow up) before day 30 were excluded from analyses. Penetrating Trauma patient population: No analysis done due to low statistical power.
Measure: Number; unit: Participants
Arm/Group | rFVIIa, Blunt Trauma | Placebo, Blunt Trauma | rFVIIa, Penetrating Trauma | Placebo, Penetrating Trauma
Number analyzed (Participants) | 218 | 242 | 0 | 0
Participants | 24 | 26 |  |
Statistical Analysis 1: Comparison: rFVIIa, Blunt Trauma vs Placebo, Blunt Trauma; Test for Odds ratio=1, corresponding to a null hypothesis of no difference in mortality for patients who died between groups for Blunt Trauma. Odds-ratio is adjusted for baseline covariates: Age, Injury Severity Score (ISS), Glasgow Coma -Scale Score (GCS), International Normalized Ratio (INR) and acute lung injury (P/F > 200). Missing covariates are imputed by the mean value; Test type: Superiority or Other; p = 0.934, Regression, Logistic — Two-sided significance level 5%
Statistical Analysis 2: Comparison: rFVIIa, Blunt Trauma vs Placebo, Blunt Trauma; Treatment groups are compared using a Cox Proportional Hazards model with treatment as factor and adjusting for age, Injury Severity Score (ISS), Glasgow Coma -Scale Score(GCS), International Normalized Ratio (INR) and acute lung injury; Test type: Superiority or Other; p = 0.589, Cox Proportional Hazards Model — Two-sided significance level 5%; Hazard Ratio (HR) = 1.18, 95% CI [0.64 to 2.17]

2. Primary Outcome: Morbidity
Description: Morbidity reflects the number of patients who had pulmonary and/or renal dysfunction requiring ongoing medical intervention on day 30.
Time Frame: from day 0 to day 30
Population: Blunt trauma patient population: According to protocol, morbidity is not part of the primary endpoint since non-inferiority test of mortality was not passed. Penetrating Trauma patient population: No analysis done due to low statistical power.
Arm/Group | rFVIIa, Blunt Trauma | Placebo, Blunt Trauma | rFVIIa, Penetrating Trauma | Placebo, Penetrating Trauma
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Days Alive and Free of Pulmonary and/or Renal Dysfunction Requiring Medical Intervention
Description: The number of days alive and free of pulmonary and/or renal dysfunction requiring medical intervention from day 0 to day 30.
Time Frame: from day 0 to day 30
Population: Blunt trauma patient population: Intention-to-treat (ITT) analysis set. Penetrating Trauma patient population: No analysis done due to low statistical power.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | rFVIIa, Blunt Trauma | Placebo, Blunt Trauma | rFVIIa, Penetrating Trauma | Placebo, Penetrating Trauma
Number analyzed (Participants) | 218 | 242 | 0 | 0
Days | 17.2 (10.3) | 16.4 (10.3) |  |
Statistical Analysis 1: Comparison: rFVIIa, Blunt Trauma vs Placebo, Blunt Trauma; Baseline covariates: Age, Injury Severity Score (ISS), Glasgow Coma -Scale Score (GCS), International Normalized Ratio (INR) and acute lung injury; Test type: Superiority or Other; p = 0.308, ANCOVA; LS means = 0.90, 95% CI [-0.83 to 2.63]

4. Secondary Outcome: Time to Death From Time of First Dose
Description: The time of first dose refers to the time of the first dose of rFVIIa or placebo.
Time Frame: from day 0 to day 30
Population: There is no measure summary for time to event type of endpoint as this would be a Kaplan-Meier graph.
Arm/Group | rFVIIa, Blunt Trauma | Placebo, Blunt Trauma | rFVIIa, Penetrating Trauma | Placebo, Penetrating Trauma
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Units of Transfused Red Blood Cells From Time of First Dose
Description: The number of units of transfused red blood cells in the first 24 hours from the time of the first dose of rFVIIa or placebo.
Time Frame: from hour 0 to 24
Population: Blunt trauma patient population: Intention-to-treat (ITT) analysis set including patients who discontinued before day 30. Penetrating Trauma patient population: No analysis done due to low statistical power.
Measure: Mean (Standard Deviation); unit: Units of transfused red blood cells
Arm/Group | rFVIIa, Blunt Trauma | Placebo, Blunt Trauma | rFVIIa, Penetrating Trauma | Placebo, Penetrating Trauma
Number analyzed (Participants) | 221 | 247 | 0 | 0
Units of transfused red blood cells | 6.9 (10.4) | 8.1 (10.9) |  |
Statistical Analysis 1: Comparison: rFVIIa, Blunt Trauma vs Placebo, Blunt Trauma; Test type: Superiority or Other; p = 0.038, Wilcoxon (Mann-Whitney); Hodges-Lehmann shift estimate = 1.0, 95% CI [0 to 2]

6. Secondary Outcome: Number of Patients Receiving 10 Units or More (Massive Transfusion) of Red Blood Cells From Time of Injury
Description: The number of patients receiving 10 units or more of red blood cells in the first 24 hours from the time of injury.
Time Frame: from hour 0 to 24
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | rFVIIa, Blunt Trauma | Placebo, Blunt Trauma | rFVIIa, Penetrating Trauma | Placebo, Penetrating Trauma
Number analyzed (Participants) | 221 | 247 | 0 | 0
Participants | 111 | 134 |  |
Statistical Analysis 1: Comparison: rFVIIa, Blunt Trauma vs Placebo, Blunt Trauma; Test type: Superiority or Other; p = 0.384, Regression, Logistic; Odds Ratio (OR) = 1.175, 95% CI [0.817 to 1.690]

7. Secondary Outcome: Number of Units of All Allogeneic Transfusions From Time of First Dose
Description: The number of units of all allogeneic transfusions in the first 24 hours from the time of the first dose of rFVIIa or placebo.
Time Frame: from hour 0 to 24
Population: Blunt trauma patient population: Intention-to-treat (ITT) analysis set, including patients who discontinued before day 30. Penetrating Trauma patient population: No analysis done due to low statistical power.
Measure: Mean (Standard Deviation); unit: Units of allogeneic transfusions
Arm/Group | rFVIIa, Blunt Trauma | Placebo, Blunt Trauma | rFVIIa, Penetrating Trauma | Placebo, Penetrating Trauma
Number analyzed (Participants) | 221 | 247 | 0 | 0
Units of allogeneic transfusions | 17.1 (26.8) | 20.7 (25.7) |  |
Statistical Analysis 1: Comparison: rFVIIa, Blunt Trauma vs Placebo, Blunt Trauma; Test type: Superiority or Other; p = 0.030, Wilcoxon (Mann-Whitney); Hodges-Lehmann shift estimate = 2, 95% CI [0 to 4]

ADVERSE EVENTS:
Time Frame: Adverse events were collected in a timespan of 90 days.
Description: Safety population includes three patients in each blunt trauma treatment arm who were randomised received an initial dose and no further information is known. These patients were not included in the intent-to-treat (ITT) population.
Arm/Group | rFVIIa, Blunt Trauma | Placebo, Blunt Trauma | rVIIa, Penetrating Trauma | Placebo, Penetrating Trauma
Serious Adverse Events (participants affected / at risk) | 147/224 | 177/250 | 18/46 | 20/40
Other Adverse Events (participants affected / at risk) | 108/224 | 125/250 | 26/46 | 24/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rFVIIa, Blunt Trauma (N=224) | Placebo, Blunt Trauma (N=250) | rVIIa, Penetrating Trauma (N=46) | Placebo, Penetrating Trauma (N=40)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 6 (6) | 8 (8) | 1 (1) | 1 (1)
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocythaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 7 (10) | 8 (9) | 2 (2) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cyanosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electromechanical dissociation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 4 (5) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperadrenalism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ulcerative keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal compartment syndrome (Gastrointestinal disorders) | 5 (5) | 7 (7) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (5) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Intestinal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal infarction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 2 (2) | 6 (6) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritoneal effusion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 10 (10) | 17 (18) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Ulcer (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound necrosis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic ischaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ischaemic hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acinetobacter infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Enterococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hepatic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incision site infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 11 (11) | 26 (27) | 3 (3) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Pseudomonas infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 24 (24) | 30 (30) | 3 (3) | 2 (2)
Septic necrosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 5 (5) | 12 (12) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skin graft infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Splenic abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Superinfection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Systemic candida (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (4) | 5 (5) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 7 (8) | 10 (10) | 0 (0) | 0 (0)
Wound infection bacterial (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Wound infection pseudomonas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound sepsis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Collapse of lung (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diffuse axonal injury (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Failure to anastomose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fat embolism (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Graft thrombosis (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hepatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Iatrogenic injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inadequate analgesia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Operative haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Traumatic liver injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary bladder rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vena cava injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weaning failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound decomposition (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac output decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sputum culture positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5) | 0 (0) | 0 (0)
Muscle necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral hygroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anoxic encephalopathy (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Brain stem haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 3 (3) | 5 (5) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Critical illness polyneuropathy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Neuromyopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraplegia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Quadriparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural effusion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope vasovagal (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 3 (3) | 3 (3) | 2 (2) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 4 (4) | 6 (6) | 0 (0) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary fistula (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 18 (18) | 0 (0) | 3 (3)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1) | 2 (2) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 7 (7) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (6) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Internal fixation of fracture (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leg amputation (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arterial thrombosis limb (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 14 (14) | 14 (14) | 0 (0) | 2 (2)
Embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Exsanguination (Vascular disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haemodynamic instability (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 5 (5) | 5 (5) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Ischaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery dissection (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 3 (3) | 6 (6) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Venous haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rFVIIa, Blunt Trauma (N=224) | Placebo, Blunt Trauma (N=250) | rVIIa, Penetrating Trauma (N=46) | Placebo, Penetrating Trauma (N=40)
Anaemia (Blood and lymphatic system disorders) | 9 (10) | 13 (14) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (10) | 15 (15) | 3 (3) | 1 (1)
Tachycardia (Cardiac disorders) | 12 (12) | 13 (14) | 6 (6) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hypothermia (General disorders) | 15 (15) | 21 (22) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 27 (27) | 27 (29) | 11 (11) | 14 (14)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 12 (12) | 17 (17) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 25 (25) | 30 (30) | 4 (4) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 28 (28) | 32 (33) | 5 (5) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 21 (21) | 28 (28) | 5 (5) | 5 (5)
Hypophosphataemia (Metabolism and nutrition disorders) | 6 (6) | 14 (14) | 4 (4) | 2 (2)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Oliguria (Renal and urinary disorders) | 9 (11) | 14 (14) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 5 (5) | 3 (3)
Hypotension (Vascular disorders) | 24 (24) | 25 (26) | 4 (4) | 4 (4)

LIMITATIONS AND CAVEATS:
Trial was terminated after planned interim analysis for futility showed a lower than expected conditional power for showing superiority (11.2% [actual] vs. 50% [required]). 554 of 1502 planned patients were included in the intent-to-treat population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk acknowledges the Investigator's right to publish the entire results of the trial in accordance with the latest Vancouver guidelines. Any such scientific paper, resentation, communication or other information concerning the investigation described in this protocol, must be submitted in writing to Novo Nordisk Trial Manager prior to submission for publication / presentation for comments. Comments will be given within four weeks from receipt of the manuscript.